CLINICAL TRIAL: NCT04966182
Title: the Application CT and MRI in the Diagnosis of Cerebral Venous Sinus Thrombosis
Brief Title: Application CT and MRI in Cerebral Venous Sinus Thrombosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-256
Record Dates: First submitted 2021-07-11; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Magnetic Resonance Imaging; Cerebral Venous Sinus Thrombosis; Computer Tomographgy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cerebral venous thrombosis (CVT) is a rare disease, and with poor prognosis. Computed tomography (CT) andmagnetic resonance imaging (MRI) are the most commonly used image modalities for patients with non-specific neurologic symptoms. We are going to assess the accuracy of CT and MRI in the differential diagnosis of CVT and cerebral venous sinus thrombosis (CVST).

ELIGIBILITY:
Inclusion Criteria:

A. The patients were diagnosed with cerebral venous thrombosis or cerebral venous sinus thrombosis; B. The patients completed at least cranial CT or MRI examination upon admission;C. The patients complete at least one of the CTV, MRV or DSA examination.

Exclusion Criteria:

A. Patients with severe cardiopulmonary insufficiency;B. Patients lost to follow-up;C. Patients with incomplete access to imaging data;D. Patients with cerebral venous sinus thrombosis that was not diagnosed at discharge.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients with the diagnosis of cerebral venous thrombosis or cerebral venous sinus thrombosis at admission were included.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
specificity and sensitivity of CT | 2022.01
  specificity and sensitivity of CT in the diagnosis of cerebral venous sinus thrombosis
specificity and sensitivity of MRI | 2022.01
  specificity and sensitivity of MRI in the diagnosis of cerebral venous sinus thrombosis

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China